CLINICAL TRIAL: NCT01754233
Title: Evaluation of the 755nm Alexandrite for the Treatment of Epidermal and Dermal Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CYN12-PICO-PL
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Dermal and Epidermal Pigmented Lesions
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite Laser (Experimental): 755nm Alexandrite Laser
  Interventions: Device: 755nm Alexandrite Laser

INTERVENTIONS:
Device: 755nm Alexandrite Laser — 755nm Alexandrite Laser for epidermal and dermal pigmented lesions

SUMMARY:
The purpose of this study is to assess treatment for facial dermal and epidermal pigmented lesions using the 755nm Alexandrite laser.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 85 years old
2. Has unwanted dermal and/or epidermal pigmented lesions or desires skin toning and wishes to undergo laser treatments.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including being photographed, following post treatment care and attending all treatment and follow up visits.
5. Has Fitzpatrick skin types III to IV.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections
4. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
5. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
6. The subject has used Accutane within 6 months prior to enrollment.
7. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
8. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
9. The subjects had prior treatment with laser or other devices in the treatment area within 3 months.
10. The subject has a history of keloids or hypertrophic scarring.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of squamous cell carcinoma or melanoma
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
14. Is allergic to topical lidocaine or topical steroids.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Photographic Evaluation | up to 4 months post last treatment

SECONDARY OUTCOMES:
Reporting of Adverse Events | up to 4 months post last treatment
Satisfaction Questionnaire | up to 4 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Skin Care Physicians, Chestnut Hill, Massachusetts, United States